CLINICAL TRIAL: NCT04466020
Title: A Self -Guided, Internet -Based Intervention for Patients With Chronic Breathlessness (SELF-BREATHE): an Interview Study.
Brief Title: SELF - BREATHE for Chronic Breathlessness
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: KCH20-056; ICA-CL-2018-04-ST2-001 (Other Grant/Funding Number: HEE/NIHR Integrated Clinical Academic Programme)
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: COPD; Cancer; Heart Failure; Interstitial Disease; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Neoplasms; Heart Failure; Dyspnea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Chronic Breathlessness: Patients with Chronic Breathlessness
  Interventions: Other: Qualitative research interviews to be conducted

INTERVENTIONS:
Other: Qualitative research interviews to be conducted — None. Qualitative research interviews to be conducted

SUMMARY:
Semi-structured qualitative interviews will be conducted to understand key factors that would enable / facilitate patients with chronic breathlessness to potentially use an online breathlessness intervention (SELF-BREATHE).

DETAILED DESCRIPTION:
STUDY OVERVIEW

Full title:

A self -guided, internet -based intervention for patients with chronic breathlessness (SELF-BREATHE): an interview study.

Objective:

To understand the key factors that would enable / facilitate patients with chronic breathlessness to use an online breathlessness support intervention (SELF-BREATHE).

Study type:

Qualitative interview study

Methods:

Semi-structured qualitative interviews will be conducted to achieve maximum variation in approx 20 patients with chronic breathlessness (a purposive sample: age sex, diagnoses, and presence of caregiver).

The interview will explore and identify:

Patients' views/experiences of internet-based activities, e.g. digital apps, shopping online; Patients' understanding, preferences, values and motivations that would influence uptake of SELF-BREATHE; Potential barriers to the development and use of SELF-BREATHE; Facilitators to usage of SELF-BREATHE, such as the ability to self-monitor progress etc...

These topics cover areas of uncertainty in order to optimise the SELF - BREATHE intervention.

Inclusion criteria:

Adult patients >18 years of age, with the ability to read, converse in English and able to provide informed consent

Chronic breathlessness on exertion and or rest (MRC dysponea score >2)

Advanced disease such as cancer, chronic obstructive pulmonary disease (COPD), chronic heart failure (CHF) or interstitial lung disease (ILD), where the underlying disease is deemed to be optimally medically managed by the referring clinician / allied health professional / clinical nurse specialist

Exclusion criteria:

Breathlessness of unknown cause

A primary diagnosis of chronic hyperventilation syndrome

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >18 years of age, with the ability to read, converse in English and able to provide informed consent
* Chronic breathlessness on exertion and or rest (MRC dyspnea score >2)
* Advanced disease such as cancer, chronic obstructive pulmonary disease (COPD), chronic heart failure (CHF) or interstitial lung disease (ILD), where the underlying disease is deemed to be optimally medically managed by the referring clinician / allied health professional / clinical nurse specialist

Exclusion Criteria:

* Breathlessness of unknown cause
* A primary diagnosis of chronic hyperventilation syndrome

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD, Cancer, Heart Failure, Interstitial Lung disease, Dyspnea
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Descriptive qualitative analysis of patients' preferences, values and motivations that would influence the use of an online self - management intervention for chronic breathlessness (SELF-BREATHE). | 12 months
  Qualitative data

CONTACTS AND LOCATIONS:
Overall Officials: Charles C Reilly, PhD,MSc,BSc, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No